CLINICAL TRIAL: NCT02204332
Title: Phase II-b Randomized Study of Cabazitaxel in Metastatic Colorectal Cancer Resistant to Standard Treatment
Brief Title: Phase II-b Randomized Clinical Trial of Cabazitaxel in Metastatic Colorectal Cancer Resistant to Standard Treatment
Acronym: COMETA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis performed on the first 10 patients showed no efficacy of cabazitaxel
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Fundación Ramón Domínguez (Other)
Responsible Party: Principal Investigator, Rafael Lopez Lopez, MD,PhD, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLL-CAB-2011-01
Record Dates: First submitted 2014-07-23; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabazitaxel (Experimental): Cabazitaxel at a dose of 25 mg / m² in a 5% dextrose or 0.9% NaCl intravenously over 1 hour, every 3 weeks (1 cycle).
  Besides, patient will be treated with BSC.
  Interventions: Drug: Cabazitaxel
- Best Supportive Care (Other): Best Supportive Care (BSC), with evaluations every 3 weeks (1 cycle).
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: Cabazitaxel
  Other Names: Jevtana
  Arms: Cabazitaxel
Other: Best Supportive Care
  Arms: Best Supportive Care

SUMMARY:
The purpose of this study is to determine efficacy and safety of cabazitaxel administration in patients with colorectal cancer resistant to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent.
* Men and women aged ≥ 18 years.
* Patients with histologically confirmed metastatic advanced colorectal cancer without the possibility of potentially curative treatment.
* Patients with a life expectancy more than three months.
* Patients with advanced colorectal cancer in progression after receiving standard treatment.
* Patients with grade 0-2 functional status, according to Eastern Cooperative Oncology Group (ECOG).
* Patients with evaluable tumor by RECIST criteria.
* Patients recovered and with a degree less than or equal to 1, or baseline of all important pre-treatment-related AEs (excluding alopecia).
* Ability and willingness of the patient to consent to participation in the study.
* Ability to understand and comply with study procedures.

Exclusion Criteria:

* Patients with a performance status greater than 2, as Eastern Cooperative Oncology Group (ECOG).
* Inadequate marrow reserve, within 7 days prior to randomization:

  * absolute neutrophil count <1.5 x 109 / L
  * Hemoglobin <9.0 g / dL
  * Platelet count <100 x 109 / L
* Inadequate liver function within 7 days prior to randomization:

  * AST (SGOT) and ALT (SGPT)> 3.0 x ULN or 5> x ULN in case of abnormal liver function due to underlying liver metastases.
  * Alkaline phosphatase> 3 × ULN (or 5 times the ULN if due to underlying liver metastases).
  * Total bilirubin> 1.5 x ULN.
* Previous history of other malignancy, except for skin basal or squamous cell cancer with proper treatment, or in situ cervical cancer, or other cancers, in which the patient has been free of the disease in the last 5 years.
* Simultaneous treatment with concomitant anticancer therapy.
* History of brain metastases, uncontrolled compression of spinal cord, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease pathologies.
* Acquired Immunodeficiency Syndrome (AIDS-related diseases) or human immunodeficiency virus (HIV) or conditions requiring antiretroviral therapy virus.
* symptomatic grade ≥ 2 peripheral sensory neuropathy, according to NCI-CTCAE v4.0.
* Any severe acute or chronic medical condition that may affect the patient's ability to participate in the study, or may lead to unacceptable security risks and non-compliance with protocol procedures or may interfere with the interpretation of the study results.
* Pregnant women or who are breastfeeding. Pregnancy assessment will be conducted by a test serum or urine during the 7 days prior to randomization.
* Patient (male or female) of reproductive age who still disagrees with the use of effective contraception during the treatment period and for at least 3 months after completion of the treatment period of the study. The definition of "effective method of birth control" is the opinion of the investigator.
* Participation in another clinical trial with an investigational drug and / or an investigational drug as adjunctive therapy within 30 days prior to randomization.
* Concomitant treatment with prohibited drugs as potent inhibitors or inducers of cytochrome P450 3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The efficacy of cabazitaxel measured by estimating the overall response rate (ORR), as the percentage of individuals who achieve a complete tumor response (CR) or partial tumor response (PR) in each arm and between arms. | From date of randomization to disease progression or until 24 months from enrolment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From randomisation to either documented disease progression or death from any cause or until 24 months from enrolment (whichever occurs earlier)

OTHER OUTCOMES:
Overall survival (OS) | From date of randomization to death from any cause or until 24 months from enrolment
Safety and toxicity in the experimental arm. Toxicity is graded according to the Common Terminology Criteria for Adverse Events (NCI-CTCAE, v 4.0). | From the date the informed consent is signed up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Rafael López López, MD, PhD, Study Chair — Hospital Clinico de Santiago
Locations (8):
- Spain (8):
  - Hospital German Trias i Pujol, Badalona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Ramón y Cajal, Madrid
  - Hospital Carlos Haya, Málaga
  - CHU de Orense, Ourense
  - Hospital Clinico de Santiago, Santiago de Compostela
  - Hospital General de Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza